CLINICAL TRIAL: NCT06123858
Title: Non-alcoholic Steatohepatitis Registry Platform Study
Status: Terminated | Type: Observational
Why Stopped: Following a reassessment of the company's pipeline priorities, the sponsor has elected to discontinue this project prior to its planned completion
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00356
Record Dates: First submitted 2023-10-25; First posted 2023-11-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: NASH With Fibrosis
Keywords: NASH；; NAFLD；; fibrosis.
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — This study plans to collect genetic information for the PNPLA3 and HSD17B13 genes from approximately 500 subjects with NASH accompanied by F2 fibrosis or higher. The genetic testing will be conducted free of charge through the blood samples collected during the screening or follow-up period and tested by a central laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NASH with fibrosis: NASH patients with fibrosis receiving routine treatment

SUMMARY:
This is a multi-center, prospective, observational registry platform study aimed at describing the clinical characteristics and diagnosis and treatment patterns of Chinese patients with nonalcoholic steatohepatitis (NASH) with fibrosis.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a metabolic stress-induced liver injury closely related to insulin resistance and genetic susceptibility, and its disease spectrum includes non-alcoholic fatty liver (NAFL), non-alcoholic steatohepatitis (NASH), cirrhosis and hepatocellular carcinoma (HCC). NASH is a severe form of NAFLD, defined as more than 5% hepatocellular steatosis combined with intralobular inflammation and hepatocellular ballooning degeneration. By conducting research on the NASH patient registry platform and collecting real-world data on the clinical characteristics and diagnosis and treatment patterns of NASH patients, including demographics, clinical characteristics, treatment, outcomes, healthcare utilization, lifestyle, and genotype, on the one hand, it can provide evidence of scientific value for clinical practice and formulate diagnosis and treatment guidelines, and on the other hand, it can promote the clinical development of NASH drugs in China.

This is a multi-center, prospective, observational registry platform study. Patient recruitment is tentatively scheduled from December 2023 to December 2024. NASH with fibrosis that meets the inclusion criteria but does not meet the exclusion criteria will be consecutively enrolled in the selected center. The estimated number of patients is 2,500, which will be adjusted according to the progress of research. Among these subjects, information on two genes, PNPLA3 and HSD17B13, will be collected from approximately 500 NASH patients with fibrosis stage F2 or higher.

ELIGIBILITY:
Inclusion Criteria:

(1) Subjects must be between 18 and 75 years old when signing the informed consent form, and must have the ability to sign the consent form independently; (2) NASH patients who meet one of the following conditions:

1. Liver biopsy was performed within 24 months before enrollment, and the pathological diagnosis was NASH and the fibrosis stage was F2 or above;
2. FibroScan-AST (FAST) score ≥ 0.30 within 24 months before enrollment;
3. There are any of the following evidences of fatty liver

   1. Controlled attenuation parameter (CAP) > 285 dB/m within 24 months before enrollment;
   2. Liver ultrasonography showed fatty liver within 24 months before enrollment;
   3. Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) examination within 24 months before enrollment showed liver fat fraction ≥ 5%; and any of the following evidence of liver fibrosis

   <!-- -->

   1. Liver stiffness measurement (LSM) ≥ 7.5kPa by vibration-controlled transient elastography (VCTE) within 24 months before enrollment;
   2. The elasticity value of magnetic resonance elastography (MRE) examination within 24 months before enrollment is ≥2.93kPa;
   3. If there is no liver biopsy and no liver elastography equipment is available in the research center, FIB-4>1.3 (under 65 years old) or>2 (over 65 years old) within 3 months before enrollment.

Exclusion Criteria:

1. History of liver transplantation;
2. Patients with bleeding tendency or coagulation dysfunction (for example, bleeding tendency, such as hemophilia, suspected hemangioma or suspected hydatid infection);
3. Exclude liver diseases caused by the following causes: alcoholic steatohepatitis, drug-induced, viral or autoimmune hepatitis, primary hemochromatosis, α1-antitrypsin deficiency, hepatolenticular degeneration, hypothyroidism, inflammatory bowel disease, Cushing's syndrome, celiac disease, β lipoprotein deficiency, lipoatrophic diabetes mellitus, Mauriac syndrome, hypopituitarism, hypogonadism, polycystic ovarian syndrome;
4. Have a history of malignant tumors in the past 5 years, excluding malignant tumors that have been cured by the investigator's judgment;
5. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with NASH and fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 1122 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
1.Patient demography | Baseline
  Gender (male, female) ，age (years)，time since pathological diagnosis of NASH (months)， proportion of comorbidities
2.The proportion of 4 NASH treatment modalities at baseline and follow-up | up to 3-year follow-up
  NASH treatment modalities include：Drug treatment，Non-drug treatment，Combined treatment and No treatment received
3.NASH Knowledge, Belief and Practice Questionnaire responses at baseline and follow-up | up to 3-year follow-up
  Describe the responses of patients to the NASH Knowledge, Belief and Practice Questionnaire at baseline and follow-up periods. The questionnaire includes NASH patients' knowledge, attitude, and behavior towards NASH disease, NASH-related medical service needs, expectations, satisfaction, and does not involve the evaluation of scores.

SECONDARY OUTCOMES:
1. The correlation between non-invasive diagnostic methods and pathological results of liver biopsy in NASH patients | up to 3-year follow-up
  Non-invasive diagnostic methods for NASH (serological or imaging indicators during baseline and follow-up periods, including FIB-4, APRI, NAFLD fibrosis score (NFS), BARD, fatty liver index (FLI), Hepatic steatosis index (HSI), VCTE, MRE, MRI-PDFF, FAST, etc.); Liver biopsy pathology: Liver biopsy pathology results during baseline and follow-up periods, including NASH pathological diagnosis, NAFLD activity score (NAS) and pathological fibrosis grade.
2.The annual frequency of liver related visits | up to 3-year follow-up
  Liver-related visits include liver related outpatient visits, emergency department visits, and hospitalizations
3.Total liver-related cost | up to 3-year follow-up
  Total liver-related cost includes total liver-related outpatient and hospitalization costs

OTHER OUTCOMES:
1.Clinical, histological and biological factors associated NASH diagnosis will be assessed using multivariate correlation | up to 3-year follow-up
  Exploring a scoring system/model for diagnosing NASH based on clinical feature data.
2.Incidence of endpoint events during follow-up period | up to 3-year follow-up
  Endpoint events include all-cause death, liver endpoint events, and extrahepatic endpoint events. Explore the risk factors for endpoint events and try to establish a prediction model for endpoint events in NASH patients.
3.Changes in Liver enzymes levels during the follow-up period compared with the baseline period | up to 3-year follow-up
  Liver enzymes assessed by alanine aminotransferase (ALT) and aspartate aminotransferase (AST)
4.Changes in the degree of steatosis during the follow-up period compared with the baseline period | up to 3-year follow-up
  Steatosis was assessed by CAP value by VCTE
5.Changes in fibrosis grades during the follow-up period compared with the baseline period | up to 3-year follow-up
  Fbrosis grade was assessed by LSM value of VCTE

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, Principal Investigator — Hepatopancreatobiliary Center, Beijing Tsinghua Changgung Hospital, Tsinghua University
Locations (16):
- China (16):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Inner Mongolia
  - Research Site, Nanchang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Xi'an
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.